CLINICAL TRIAL: NCT00975832
Title: Adipose Expression of Leptin, Adiponectin and IL-6, and Plasma Levels of Adipocytokines in Lean and Obese Women With PCOS
Brief Title: Adipocytokines and Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Statens Serum Institut (Other); Aarhus University Hospital (Other)
Responsible Party: Pernille Fog Svendsen, MD, Copenhagen University Hospital, Hvidovre
Other Study IDs: PSvendsen
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: The independent effect of PCOS and obesity on adipose expression and plasma levels of adipocytokines
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- women with polycystic ovary syndrome
- women without polycystic ovary syndrome
- women from 18-40 years of age

SUMMARY:
Inflammation may play a role in the development of polycystic ovary syndrome (PCOS). In this study, the investigators investigated the expression of different mediators of inflammation in fatty tissue and in blood in women with and without PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS were included according to the Rotterdam diagnostic criteria for PCOS. Control women met none of the criteria for PCOS

Exclusion Criteria:

* Oc´s within the last three months, or other medication known to alter glucose/insulin metabolism
* Other known chronic diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 36 women (17 lean and 19 obese)with PCOS and 24 (8 lean and 16 obese) control women
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)

REFERENCES:
- [Derived] Svendsen PF, Christiansen M, Hedley PL, Nilas L, Pedersen SB, Madsbad S. Adipose expression of adipocytokines in women with polycystic ovary syndrome. Fertil Steril. 2012 Jul;98(1):235-41. doi: 10.1016/j.fertnstert.2012.03.056. Epub 2012 May 16. PMID 22607892